CLINICAL TRIAL: NCT04688320
Title: Multicenter, Open Label, Randomized Comparative Trial of the Efficacy and Safety of a Single Bolus Recombinant Non-immunogenic Staphylokinase and Bolus-infusion of Alteplase in Patients With Massive Pulmonary Embolism (FORPE)
Brief Title: Massive Pulmonary Embolism: Trial of Non-immunogenic Recombinant Staphylokinase VS Alteplase FORPE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Supergene, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FORPE
Record Dates: First submitted 2020-12-18; First posted 2020-12-29 (Actual); Results first posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Massive Pulmonary Embolism
Keywords: Massive pulmonary embolism; Fibrinolysis; Recombinant Non-immunogenic Staphylokinase
MeSH Terms: interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Intervention Model Description: At clinical centers, patients will be equally randomly distributed by the "envelope method" into two groups to receive Fortelizin® or Alteplase®.
  The drugs will be administered after the signed informed consent. Fortelizin® will be administered intravenously at a dose of 15 mg as a single bolus for 10-15 seconds. Alteplase® will be administered in accordance with the instructions for use. All patients will be examination for 30 days.
Masking Description: All eligible patients will be randomized in two equal groups for administration recombinant nonimmunogenic staphylokinase (Fortelyzin) or alteplase (Actilize) by using "envelope method" of randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant nonimmunogenic staphylokinase (Experimental): lyophilisate for preparation of a solution for intravenous administration, 5 mg (745,000 IU) complete with a solvent. 15 mg (2,235,000 IU) - 3 vials, intravenously as a quick single bolus injection for 10-15 seconds, regardless of body weight.
  Interventions: Drug: Recombinant nonimmunogenic staphylokinase
- Alteplase (Experimental): Alteplase® is administered in accordance with the instructions for use for pulmonary embolism( 10 mg bolus and 90 mg as IV infusion over 2 hours, maximum 100 mg). In patients weighing less than 65 kg, the total dose should not exceed 1.5 mg / kg.
  Interventions: Drug: Alteplase

INTERVENTIONS:
Drug: Recombinant nonimmunogenic staphylokinase — 15 mg of drug reconstituted in 10 ml of 0.9% solution of NaCl given as single i.v. bolus over 10-15 seconds
  Other Names: Fortelyzin
  Arms: Recombinant nonimmunogenic staphylokinase
Drug: Alteplase — Alteplase® is administered in accordance with the instructions for use for pulmonary embolism ( 10 mg bolus and 90 mg as IV infusion over 2 hours, maximum 100 mg). In patients weighing less than 65 kg, the total dose should not exceed 1.5 mg / kg.
  Other Names: Actillyze
  Arms: Alteplase

SUMMARY:
Objective: to evaluate the efficacy and safety of the Recombinant Non-immunogenic Staphylokinase with its single bolus administration in comparison with the bolus-infusion administration of the Alteplase in patients with massive pulmonary embolism

DETAILED DESCRIPTION:
The main goal of treating massive PE is to save the lives of patients by restoring pulmonary perfusion, preventing the development of chronic postembolic pulmonary hypertension and recurrent PE. According to data of clinical trials, with timely initiation of therapy for massive pulmonary embolism, mortality can be significantly reduced.

Recombinant protein which contains aminoacid sequence of staphylokinase - Fortelizin® (the active substance is Forteplase). It is single chain molecula, consists of 138 aminoacids, weight 15.5 kDa. When staphylokinase is added to human plasma containing a fibrin clot, it preferentially reacts with plasmin at the clot surface, forming a plasmin-staphylokinase complex. This complex activates plasminogen trapped in the thrombus. The plasmin-staphylokinase complex and plasmin bound to fibrin are protected from inhibition by alpha2-antiplasmin. Once liberated from the clot (or generated in plasma), however, they are rapidly inhibited by alpha2-antiplasmin. This selectivity of action confines the process of plasminogen activation to the thrombus, preventing excessive plasmin generation, alpha2-antiplasmin depletion, and fibrinogen degradation in plasma. In rabbits anti forteplase antibodies are not produced. It was achieved by replacement of amino acids in immunogenic epitop of molecule staphylokinase. Blood fibrinogen decrease after i.v. injection of Fortelyzin less 10% within first 24 hours. Angiographic data suggests that restoration of coronary blood flow appears in up to 80% of patients with STEMI after i.v. injection of Fortelyzin.

The main objectives of the study: to assess the efficacy, safety and possible adverse events of the drug Recombinant Non-immunogenic Staphylokinase with its single bolus administration in comparison with the bolus-infusion administration of the drug Alteplase® in patients with massive pulmonary embolism.

Study Design. Multicenter, open-label, randomized, comparative clinical study of non-inferiority study of efficacy and safety in parallel groups. At clinical centers, patients will be equally randomly distributed by the "envelope" method into two groups of 155 patients each (310 people in total, including 10% of those who may have dropped out)to receive Recombinant Non-immunogenic Staphylokinase or Alteplase®.

The drugs will be administered after the signed informed consent. Recombinant Non-immunogenic Staphylokinase will be administered intravenously at a dose of 15 mg as a single bolus for 10-15 seconds. Alteplase® will be administered in accordance with the instructions for use.

Patients will be monitored for 30 days from the moment of randomization: in the intensive care unit up to 7 days, after it in the hospital until discharge - an average of 14 days and an outpatient visits on the 30th day. The recruitment of patients for the study will be competitive.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 and over
* Verified diagnosis of massive PE (using MSCT with PA contrast)
* Signs of overload / dysfunction of the right ventricle (at least one) in combination with persistent arterial hypotension or shock
* Patient consent to use reliable contraceptive methods throughout the study and for 3 weeks after:

  * women who have a negative pregnancy test and use the following contraceptives: intrauterine devices, oral contraceptives, contraceptive patch, prolonged injectable contraceptives, double barrier method of contraception. Women who are not fertile can also take part in the study (documented conditions: hysterectomy, tubal ligation, infertility, menopause for more than 1 year);
  * men using barrier contraception. The study may also involve men who are not fertile (documented conditions: vasectomy, infertility)
* Availability of signed and dated informed consent of the patient to participate in the study.

Exclusion Criteria:

* • Increased risk of bleeding:

  * Extensive bleeding at present or within the previous 6 months, hemorrhagic diathesis;
  * Intracranial (including subarachnoid) hemorrhage at present or in history, suspected hemorrhagic stroke;
  * A history of hemorrhagic stroke or stroke of unknown etiology;
  * Ischemic stroke or transient ischemic attack within the last 6 months, except for the current acute ischemic stroke within 4.5 hours;
  * A history of diseases of the central nervous system (including neoplasms, aneurysms, surgery on the brain or spinal cord);
  * Major surgery or major trauma within the previous 3 months, recent traumatic brain injury;
  * Long-term or traumatic cardiopulmonary resuscitation (> 2 min), delivery within the previous 10 days, recent puncture of an uncompressible blood vessel (eg, subclavian or jugular vein);
  * Severe liver disease, including liver failure, cirrhosis, portal hypertension (including esophageal varices) and active hepatitis;
  * Confirmed gastric or duodenal ulcer within the last three months;
  * Neoplasm with an increased risk of bleeding;
  * Concurrent administration of oral anticoagulants, for example, warfarin with an INR> 1.3;
  * Arterial aneurysms, developmental defects of arteries / veins;
  * Severe uncontrolled arterial hypertension;
  * Acute pancreatitis;
  * Bacterial endocarditis, pericarditis;
  * suspicion of aortic dissecting aneurysm;
  * any other conditions, in the opinion of the doctor, associated with a high risk of bleeding.
* Lactation, pregnancy
* Known hypersensitivity to Alteplase, Fortelizin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander I Kirienko, MD, PhD, Principal Investigator — Pirogov Russian National Research Medical University; Sergey S Markin, MD, PhD, Study Director — Supergene, LLC
Locations (23):
- Russia (23):
  - V.F. Dolgopolov Vyselki Central District Hospital, Vyselki, Krasnodarskiy Kray
  - Sergiyev Posad Regional Clinical Hospital, Sergiyev Posad, Moscow Oblast
  - Belgorod Regional Clinical Hospital of St. Joseph, Belgorod
  - Kuzbass Cardiology center, Kemerovo
  - Krasnoyarsk Regional Clinical Hospital, Krasnoyarsk
  - Kursk Regional Clinical Hospital, Kursk
  - D.D. Pletnev City Clinical Hospital, Moscow
  - I.V. Davydovskii City Clinical Hospital, Moscow
  - S.S. Yudin City Clinical Hospital, Moscow
  - V.V. Vinogradov City Clinical Hospital, Moscow
  - V.V. Veresaev City Clinical Hospital, Moscow
  - N.V. Sklifosovsky Research Institute for Emergency Medicine, Moscow
  - S.P. Botkin City Clinical Hospital, Moscow
  - Murmansk Regional Clinical Hospital, Murmansk
  - N.N. Burdenko Penza Regional Clinical hospital, Penza
  - G.A. Zakharyin Clinical hospital №6, Penza
  - Saint Petersburg "Mariinskaya" City Hospital, Saint Petersburg
  - Holy Martyr Elizabeth Saint Petersburg City Hospital, Saint Petersburg
  - V.P. Polyakov Samara Regional Clinical Cardiology Dispensary, Samara
  - Saratov Regional Clinical Cardiology Dispensary, Saratov
  - Tver Regional Clinical Hospital, Tver'
  - City Clinical hospital №4, Vladimir
  - City Clinical Hospital of Emergency №25, Volgograd

REFERENCES:
- [Derived] Leontyev SG, Yarovaya EB, Kutsenko VA, Ivlev OE, Soplenkova AG, Semenov AM, Semenov MP, Ivanov SV, Romashova YA, Markin SS. The Safety of Non-immunogenic Recombinant Staphylokinase in Elderly Patients With Massive Pulmonary Embolism: A Randomized Clinical Trial FORPE. Health Sci Rep. 2025 May 19;8(5):e70826. doi: 10.1002/hsr2.70826. eCollection 2025 May. PMID 40391253

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Recombinant Nonimmunogenic Staphylokinase | Alteplase
Started | 155 | 155
Completed | 145 | 146
Not Completed | 10 | 9

BASELINE CHARACTERISTICS:
Population: 310 patients were randomly assigned to receive either non-immunogenic staphylokinase (n=155) or alteplase (n=155)
Groups:
- Total: Total of all reporting groups
Arm/Group | Recombinant Nonimmunogenic Staphylokinase | Alteplase | Total
Number analyzed (Participants) | 155 | 155 | 310
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 75 | 94 | 169
  >=65 years | 80 | 61 | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (13) | 62 (13) | 63 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 74 | 158
  Male | 71 | 81 | 152
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 155 | 155 | 310
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russia | 155 | 155 | 310
Body mass index, kg/m^2 [Mean (Standard Deviation); unit: kg/m^2] | 32 (6) | 31 (6) | 32 (6)
Pulmonary Embolism Severity Index (PESI) score [Median (Inter-Quartile Range); unit: score] — Pulmonary embolism severity index (PESI). PESI evaluates the patient's age and mortality risk factors. The minimum score on the PESI scale = the patient's age, the maximum = the patient's age + 230 points. If total PESI score is ≤ 65, patient has a very low risk of mortality; 66-85 score - a low risk of mortality; 86-105 score - an intermediate risk of mortality; 106-125 score - a high risk of mortality; if PESI score > 125, patient has a very high risk of mortality.
  score | 135 [116 to 150] | 128 [113 to 145] | 132 [115 to 147]
PESI class V patients [Count of Participants; unit: Participants] — Patients, who have pulmonary embolism severity index (PESI) > 125 score, considered as a class V, with a very high risk of mortality
  Participants | 103 | 82 | 185
Onset to treatment time [Median (Inter-Quartile Range); unit: h] | 27 [11.8 to 80.5] | 17.1 [8.5 to 68.5] | 22 [9.2 to 72.5]
Qanadli index [Mean (Standard Deviation); unit: % of pulmonary artery obstruction] — To quantify the degree of pulmonary artery obstruction by CTPA, the Qanadli index was calculated, where 0 points means no obstruction, 40 points means complete occlusion of all branches of the pulmonary artery.
  The percentage (%) of pulmonary artery obstruction was calculated by dividing the patient's score by the maximum score (40) and and multiplying the result by 100.
  % of pulmonary artery obstruction | 65.8 (19.8) | 67.8 (19.7) | 66.2 (19.8)
Right ventricle end-diastolic diameter [Median (Inter-Quartile Range); unit: mm] | 50 [45 to 56] | 50 [47 to 55] | 50 [46 to 56]
Right ventricular/lLeft ventricular end-diastolic diameter [Median (Inter-Quartile Range); unit: ratio] — Ratio of right ventricular (RV) end-diastolic diameter to left ventricular (LV) end-diastolic diameter
  ratio | 1.39 [1.30 to 1.52] | 1.40 [1.34 to 1.51] | 1.40 [1.32 to 1.52]
Baseline systolic blood pressure [Median (Inter-Quartile Range); unit: mm Hg] | 90 [85 to 100] | 90 [85 to 100] | 90 [85 to 100]
Baseline diastolic blood pressure [Median (Inter-Quartile Range); unit: mm Hg] | 60 [52 to 65] | 60 [53 to 69] | 60 [53 to 67]
Baseline heart rate [Median (Inter-Quartile Range); unit: beats per min] | 110 [90 to 115] | 110 [92 to 115] | 110 [91 to 115]
Baseline respiratory rate [Median (Inter-Quartile Range); unit: breaths per min] | 24 [20 to 27] | 24 [21 to 26] | 24 [21 to 27]
Baseline SpO2 [Median (Inter-Quartile Range); unit: %] | 89 [88 to 90] | 89 [88 to 92] | 89 [88 to 91]

OUTCOME MEASURES:

1. Primary Outcome: Death From All Causes
Description: The efficacy is evaluated in terms of the number of deaths from all causes
Time Frame: within 7 days
Population: in the per-protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant Nonimmunogenic Staphylokinase | Alteplase
Number analyzed (Participants) | 145 | 146
Participants | 3 | 4
Statistical Analysis 1: Comparison: Recombinant Nonimmunogenic Staphylokinase vs Alteplase; Test type: Non-Inferiority — The margin of the non-inferiority was established as a difference in the primary efficacy endpoints between compared groups; p < 0.05, Welch's t-test; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.11 to 4.52]

2. Secondary Outcome: Systolic Pulmonary Artery Pressure Measures (V1, V2, V4, V5)
Description: The efficacy is evaluated in terms of systolic pulmonary artery pressure values
Time Frame: baseline and day 1, 7, 14 after randomisation
Population: The efficacy is evaluated in terms of decreasing of pulmonary artery systolic pressure (PASP) values on baseline and day 1, 7, 14 after randomisation in the per-protocol population
Measure: Median (Inter-Quartile Range); unit: mm Hg
Arm/Group | Recombinant Nonimmunogenic Staphylokinase | Alteplase
Number analyzed (Participants) | 145 | 145
mm Hg
  PASP on baseline | 59 [50 to 69] | 58 [51 to 69]
  PASP on day 1 | 44 [36 to 52] | 42 [36 to 50]
  PASP on day 7 | 36 [31 to 44] | 35 [29 to 41]
  PASP on day 14 | 35 [30 to 41] | 35 [28 to 41]

3. Secondary Outcome: Haemodynamic Collapse
Description: The efficacy is evaluated in terms of the number of haemodynamic collapse
Time Frame: within 7 days
Population: The efficacy is evaluated in terms of the number of haemodynamic collapse in the per-protocol population
Measure: Number; unit: events
Arm/Group | Recombinant Nonimmunogenic Staphylokinase | Alteplase
Number analyzed (Participants) | 145 | 146
events | 1 | 3

4. Secondary Outcome: Recurrent Pulmonary Embolism (PE)
Description: The efficacy is evaluated in terms of the number of recurrent PE
Time Frame: within 7 days
Population: The efficacy is evaluated in terms of the number of recurrent PE in the per-protocol population
Measure: Number; unit: events
Arm/Group | Recombinant Nonimmunogenic Staphylokinase | Alteplase
Number analyzed (Participants) | 145 | 146
events | 1 | 2

5. Secondary Outcome: Death From PE
Description: The efficacy is evaluated in terms of the number of deaths from PE
Time Frame: within 30 days
Population: The efficacy is evaluated in terms of the number of deaths from PE in the per-protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant Nonimmunogenic Staphylokinase | Alteplase
Number analyzed (Participants) | 145 | 146
Participants | 4 | 2

6. Secondary Outcome: Death From All Causes
Description: The efficacy is evaluated in terms of the number of deaths from all causes
Time Frame: within 30 days
Population: The efficacy is evaluated in terms of the number of deaths from all causes in the per-protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant Nonimmunogenic Staphylokinase | Alteplase
Number analyzed (Participants) | 145 | 146
Participants | 6 | 4

7. Secondary Outcome: Haemodynamic Collapse Within 7 Days + Recurrent PE Within 7 Days + Death From All Causes Within 30 Days
Description: The efficacy is evaluated in terms of the number of haemodynamic collapse + recurrent PE + deaths from all causes
Time Frame: within 30 days
Population: The efficacy is evaluated in terms of the number of haemodynamic collapse + recurrent PE + deaths from all causes within 30 days in the per-protocol population
Measure: Number; unit: events
Arm/Group | Recombinant Nonimmunogenic Staphylokinase | Alteplase
Number analyzed (Participants) | 145 | 146
events | 8 | 9

8. Secondary Outcome: Safety Endpoint - Haemorrhagic Stroke
Description: The safety is evaluated in terms of the number of haemorrhagic stroke within 7 days of randomisation
Time Frame: within 7 days
Population: The safety is evaluated in terms of the number of haemorrhagic stroke within 7 days of randomisation in the per-protocol population
Measure: Number; unit: events
Arm/Group | Recombinant Nonimmunogenic Staphylokinase | Alteplase
Number analyzed (Participants) | 145 | 146
events | 0 | 3

9. Secondary Outcome: Safety Endpoint - BARC Type 3+5 Bleeding
Description: The safety is evaluated in terms of the number of BARC type 3+5 bleeding. Type 3a: overt bleeding plus a hemoglobin drop of 3 to 5 g/dL; any transfusion with overt bleeding.
  Type 3b: overt bleeding plus a hemoglobin drop of 5 g/dL; cardiac tamponade; bleeding requiring surgical intervention for control; bleeding requiring intravenous vasoactive agents.
  Type 3c: intracranial hemorrhage (does not include microbleeds or hemorrhagic transformation, does include intraspinal); subcategories confirmed by autopsy or imaging, or lumbar puncture; intraocular bleed compromising vision.
  Type 5a: probable fatal bleeding; no autopsy or imaging confirmation but clinically suspicious.
  Type 5b: definite fatal bleeding; overt bleeding or autopsy, or imaging confirmation.
Time Frame: within 30 days
Population: The safety is evaluated in terms of the number of BARC type 3+5 bleeding within 30 days in the per-protocol population
Measure: Number; unit: events
Arm/Group | Recombinant Nonimmunogenic Staphylokinase | Alteplase
Number analyzed (Participants) | 145 | 146
events | 0 | 5

10. Secondary Outcome: Safety Endpoint - Number and Severity of Serious Adverse Events (SAEs)
Description: The safety is evaluated in terms of the number and severity of serious adverse events (SAEs)
Time Frame: within 30 days
Population: The safety is evaluated in terms of the number and severity of serious adverse events (SAEs) in the per-protocol population
Measure: Number; unit: events
Arm/Group | Recombinant Nonimmunogenic Staphylokinase | Alteplase
Number analyzed (Participants) | 145 | 146
events | 9 | 17

ADVERSE EVENTS:
Time Frame: 30 days.
Description: Death from all causes; Recurrent PE; Haemodynamic collapse; Ischaemic stroke; Haemorrhagic stroke; Cerebral oedema; Brainstem damage; Haematoma of the thigh; Pulmonary haemorrhage.
Arm/Group | Recombinant Nonimmunogenic Staphylokinase | Alteplase
All-Cause Mortality (participants affected / at risk) | 6/145 | 4/146
Serious Adverse Events (participants affected / at risk) | 9/145 | 17/146
Other Adverse Events (participants affected / at risk) | 72/155 | 86/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Nonimmunogenic Staphylokinase (N=145) | Alteplase (N=146)
Recurrent PE (Cardiac disorders) | 1 (1) | 2 (2) — 30 days
Haemodynamic collapse (Cardiac disorders) | 1 (1) | 3 (3) — 30 days
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) — 30 days
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 3 (3) — 30 days
Cerebral oedema (Nervous system disorders) | 0 (0) | 2 (2) — 30 days
Brainstem damage (Nervous system disorders) | 0 (0) | 1 (1) — 30 days
Haematoma of the thigh (Cardiac disorders) | 0 (0) | 1 (1) — 30 days
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — 30 days
Death from all causes (Cardiac disorders) | 6 (6) | 4 (4) — 30 days
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Nonimmunogenic Staphylokinase (N=155) | Alteplase (N=155)
Hematuria (Blood and lymphatic system disorders) | 72 (72) | 86 (86)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT04688320/Prot_SAP_000.pdf
  • Informed Consent Form (2018-09-01): https://cdn.clinicaltrials.gov/large-docs/20/NCT04688320/ICF_001.pdf